CLINICAL TRIAL: NCT03546920
Title: Integrating Palliative Care Social Workers Into Sub-Acute Settings: A Feasibility Trial
Acronym: ALIGN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Kaiser Permanente (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: 17-2263
Record Dates: First submitted 2018-05-23; First posted 2018-06-06 (Actual); Last update posted 2019-07-10 (Actual); Status verified 2019-07

CONDITIONS: Advanced Medical Illness

STUDY DESIGN:
Intervention Model Description: Step wedge design. Randomization occurred at the facility level. Facilities are randomized to the order of starting accrual in control phase and then transitioning to intervention phase once control sample has accrued.
Masking Description: This is a feasibility trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Phase (No Intervention): Usual care for patients admitted to the SNF.
- ALIGN Intervention Phase (Experimental): ALIGN Intervention delivered by Palliative Care Social Workers in the SNF setting. The intervention consists of aligning patient/caregiver goals of care, completing advance care planning, and connecting to community resources and services to ensure smooth transition from facility to home setting.
  Interventions: Behavioral: ALIGN Intervention Phase

INTERVENTIONS:
Behavioral: ALIGN Intervention Phase — Communication: The PCSW will follow this structured process to improve and facilitate communication for intervention patients. 1. Attend routine weekly facility-led rounds/meetings reviewing patients, their needs and attend discharge planning conference; 2. Visit with patient and caregiver after the discharge planning conference to ensure understanding of the plan of care; 3. Ensure all appropriate community programs (home health, community palliative care) have made contact and established care, assess the transition, and revisit domains from the initial assessment; 4. Suggest questions that need to be asked of community providers. Throughout the intervention, the PCSW will communicate updates from the visits to all involved providers.
  Visits will also focus on increasing goal alignment with the objective that all participants have a ROLT score that is most aligned. Visits will also explore goals of care; this includes completion or review of advance directives.
  Arms: ALIGN Intervention Phase

SUMMARY:
This is a feasibility trial utilizing a step wedge design of a social worker led palliative care intervention for 120 adult patients with advanced medical illness being cared for in a subacute nursing facility. Caregivers are also invited to participate.

DETAILED DESCRIPTION:
Of the nearly 800,000 seniors admitted to Skilled Nursing Facilities for rehabilitation (SNF rehab) annually in the U.S., approximately 20% will be newly institutionalized, 25-50% are readmitted back to the hospital within 30 days at a cost of $4.34 billion, and 9% will die in the next year. Clearly this population represents an ideal target for palliative care interventions such as decreasing symptom burden, improving quality of life, and ensuring that the medical care provided is congruent with patient goals and preferences. Unfortunately, health professionals working in the SNF rehab setting are rarely trained in palliative care. While the current standard of care in the SNF rehab setting typically includes social service assessment and case management, the care plans developed are frequently focused only on immediate, short-term issues and are not communicated as the patient is discharged to a different level of care. Existing literature supports the need to assist patients in navigating care transitions through standardized systems and patient/family activation. However, the transition from hospital to SNF and from SNF to community has received little attention, even though these are some of the most complex patients at high risk for poor outcomes. The broad goal of the research team is to optimize care for high-risk seniors admitted to SNF rehab by using a social work led, therapeutic intervention designed to align goals of care and improve communication across multiple care settings.

ALIGN (Assessing & Listening to Individual Goals and Needs), a palliative social work led intervention, focuses on defining patient and caregiver goals and values through an ecological assessment with standardized monitoring and reassessment, providing education about disease trajectory, facilitating communication between the patient and the care team, and developing a patient-centered care plan that accompanies the patient across all future transitions. ALIGN was previously tested in a long-term acute care hospital setting as part of a quality improvement project that demonstrated decreased hospital readmissions, increased use of hospice, improved self-reported patient care experience, and higher levels of advance directive completion. This pilot study will be conducted to determine the feasibility of applying ALIGN to the SNF rehab population. The current protocol will enroll 60 patients aged 65+ at the time of admission to receive the ALIGN intervention along with at least 60 caregivers. The Investigators will also enroll 120 patients and 60 caregivers to receive care as usual. The proposed specific aims (SA) and Hypotheses (H) are:

SA1: To determine the feasibility of conducting a trial of ALIGN in older persons and their caregivers admitted to SNF rehab using a pragmatic, stepped-wedge design.

H1: The ALIGN intervention will be feasible if a) eligibility, enrollment, refusal, retention and attrition rates are within 20% of expected; b) facility staff/providers and participants (patients and caregivers) find the intervention acceptable (semi-structured qualitative interviews)

SA2: To conduct an exploratory analysis to estimate the effect size of ALIGN vs usual care on the primary patient-centered outcome, quality of life (FACT-G), and caregiver-centered outcome, caregiver burden (Zarit caregiver burden scale) and the secondary outcome (health care utilization). The investigators hypothesize that compared to control at 60-days post-enrollment, the ALIGN subjects will have:

H2a: A clinically meaningful difference in the FACT-G (3-7 points on the overall scale) for patients.

H2b: A clinically meaningful difference in the Zarit Caregiver burden scale (8±15) for caregivers.

H2c: A 20% relative decrease in 60-day readmission to hospital.

In addition to the key primary and secondary outcome measures listed above, the investigators will also explore the effect of ALIGN on utilization of palliative care/hospice, hospital length of stay, advance directive documentation, and care experience (Advanced Illness Coordinating Care Survey).

ELIGIBILITY:
Inclusion Criteria:

High risk for hospital readmission based on LACE Score > 7;

* Length of stay in days,
* Caregivers must be > 18 years old,
* Comorbidity,
* ER Visits in past 6 months)
* Admitted to SNF
* Decisional capacity to consent or proxy available to consent
* English speaking

Exclusion Criteria:

* Lacking proxy available for consent

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 220 (Actual)
Dates: Start 2018-01-08 (Actual); Primary Completion 2019-06-16 (Actual); Study Completion 2019-06-16 (Actual)

PRIMARY OUTCOMES:
Feasibility | 60 days
  Number approached, enrolled, and retained in the collection of patient reported outcome measures

SECONDARY OUTCOMES:
Change in Quality of Life | Baseline and 60 days
  FACT-G
Change in Caregiver Reaction Assessment | Baseline and 60 days
  Caregiver burden and benefit finding
Change in Zarit Caregiver Burden | Baseline and 60 days
  burdens of caregiving
Change in AICCES Survey | Baseline and 60 days
  A survey of satisfaction with care for patients and caregivers

CONTACTS AND LOCATIONS:
Overall Officials: Stacy M Fischer, MD, Principal Investigator — University of Colorado SOM
Locations (1):
- Kaiser Permanente Colorado-N/S/W, Denver, Colorado, United States

IPD SHARING:
Plan to Share IPD: No
No plan to share IPD outside research team